CLINICAL TRIAL: NCT06952218
Title: Effect of Cross-linked Hyaluronic Acid Filler Versus Botulinum Toxin Type A (Botox) in Management of Gummy Smile: Randomized Controlled Clinical Trial
Brief Title: Effect of Cross-linked Hyaluronic Acid Filler Versus Botulinum Toxin Type A (Botox) in Management of Gummy Smile
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Raghda Hussein Metwaly Mahmoud, Masters Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5699269
Record Dates: First submitted 2025-04-15; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Gummy Smile Due to Hypermobile Upper Lip

STUDY DESIGN:
Intervention Model Description: Lidocaine 5% ointment will be applied to the intended injection site for 20 mins. In control group, 2.5 units of botulinum toxin will be injected bilaterally at Yonsei Point. An insulin needle will be used for injecting the botox. In intervention group, a bolus of 0.2 ml of 20% cross linked hyaluronic acid filler will be injected in canine fossa region using a 29G needle preceeded by aspiration for 10 seconds ensuring no blood vessel will be involved. The product will be infiltrated slowly keeping an angle of 90 degrees in relation to the bone.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I will receive botulinum toxin type A injection. (Active Comparator): Injection site will be determined at a point in which the elevator muscles of the upper lip which are levator labii superioris, levator labii superioris alaeque nasi, and zygomaticus minor converge into the lateral area of the ala of the nose. The center of intersection of the mentioned muscles is termed Yonsei Point and estimated to be at a 1cm horizontal distance from the ala of the nose and a 3cm vertical distance from the lip line. Lidocaine 5% ointment will be applied to the intended injection site for 20 mins. In control group, 2.5 units of botulinum toxin will be injected bilaterally at Yonsei Point. An insulin needle will be used for injecting the botox.
  Interventions: Procedure: Injection of cross linked hyaluronic acid filler
- Group II will receive cross linked hyaluronic acid filler injection (Experimental): Lidocaine 5% ointment will be applied to the intended injection site for 20 mins. In intervention group, a bolus of 0.2 ml of 20% cross linked hyaluronic acid filler will be injected in canine fossa region using a 29G needle preceeded by aspiration for 10 seconds ensuring no blood vessel will be involved.
  Interventions: Procedure: Injection of cross linked hyaluronic acid filler

INTERVENTIONS:
Procedure: Injection of cross linked hyaluronic acid filler — Injection of cross linked hyaluronic acid filler

SUMMARY:
A smile is supposed to express one's feelings and expressions, for that there has been an awakening concern for the appearance of gummy smile. Gummy smile is the appearance of about 2mm or more of the gingiva during smiling. It may affect the quality of life of individuals affecting their self-esteem; patients desire to look good not only while resting but while dynamically expressing themselves too. Variable factors contribute to this gingival display whether skeletal, dental or muscular. Variable treatment modalities are done solely or in adjunction to each other for the treatment of gummy smile including both surgical or nonsurgical procedures.

DETAILED DESCRIPTION:
In patients not preferring surgical correction of gummy smile, botulinum toxin injection type A can be a helpful solution for reduction of peri-oral muscular hypermobility. A characteristic feature of botulinum toxin is the need for the re-injection in short intervals of time to yield better lasting effects. The use of cross-linked hyaluronic acid dermal fillers when used to myomodulate the peri-oral muscles give more immediate results and reduces the need for re-injection at shorter intervals.

Botulinum toxin type A, a toxin produced by the bacteria Clostridium botulinum, has been widely used in different therapeutic and cosmetic applications in dentistry. Amongst its important applications is the treatment of gummy smile by reducing the hypermobility of the peri-oral muscles through chemical denervation. Botox elicits temporary results and requires re-injection at certain time points. It is a safe, suitable, transient solution for patients not willing to undergo any surgical intervention to manage their gummy smile. Another approach for the non invasive treatment of muscular hypermobility is the injection of cross linked hyaluronic acid filler. Once the filler is injected, it typically occupies space that lessens the muscle movement limiting its hypermobility. Instant Smile enhancement is observed upon injection of cross-linked hyaluronic acid fillers and no need to repeat the injection at closer periods of time. Hyaluronic acid fillers are non-permanent fillers that are degradable by hyaluronidase and cross linking renders them more resistant to enzymatic degradation thus lasting longer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with excessive gingival display ranging from 3-8mm due to hypermobile lip.
* Age ranges from 18 years or above.

Exclusion Criteria:

* Excessive gingival display due to other etiological factors.
* Patients allergic to botox or hyaluronic acid fillers.
* Patients with any medical condition that contraindicates botox or hyaluronic acid filler injection.
* Patients previously injected with permanent fillers.
* Pregnancy.
* Breastfeeding females.
* Patients with active inflammatory or infectious disease at intended site of injection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Gingival display | week 2, month 1, month 3, month 6, month 9
  will be measured from a point denoting the lowest margin of the upper lip perpendicular and superior to the midportion of the gingival margin of the maxillary lateral incisor to the gingival margin at the midpoint of the maxillary lateral incisor.
  The midpoint of the incisal edge of the maxillary lateral incisor will be used as a reference point if the upper lip fell below the gingival margin of the same tooth post-injection (Diaspro, Cavallini et al. 2018).

SECONDARY OUTCOMES:
Patient satisfaction | week 2, month 1, month 3, month 6, month 9
  The patient will be asked to rate the satisfaction about her/his smile on a scale from 1 to 5 where 1 represents the least satisfied and 5 indicates the most (Makkeiah, Harfoush et al. 2021).
Postoperative pain | week 2, month 1, month 3, month 6, month 9
  The patient will be asked to mark her/his current level of pain on a scale of 10 cm line denoting a range between zero being (no pain) to 10 (maximum pain) (Diaspro, Cavallini et al. 2018).
Lip mobility | week 2, month 1, month 3, month 6, month 9
  will be measured by subtracting upper lip length during smiling from upper lip length at rest (Sabbah 2022). The upper lip length is measured from the subnasale to the lower border of the upper lip at the central incisors' region at smile and rest (Ali, Kilani et al. 2023).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - CairoU, Cairo
  - Cairo University, Giza

IPD SHARING:
Plan to Share IPD: No